CLINICAL TRIAL: NCT04985396
Title: Effect of Platelet Rich Plasma Injection Compared With Steroid Injection for the Treatment of Plantar Fasciitis: A Randomized Clinical Trial
Brief Title: Platelet Rich Plasma Injection Compared With Steroid Injection for the Treatment of Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Police Force Hospital, Nepal (Other Government)
Responsible Party: Principal Investigator, Dev Ram Sunuwar, Assistant Professor, Armed Police Force Hospital, Nepal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plantar Fasciitis
Record Dates: First submitted 2021-07-14; First posted 2021-08-02 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Plantar Fasciitis; Steroid; Platelet-rich Plasma (PRP)
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: A hospital-based randomized clinical trial study will be carried out to compare the efficacy of steroid injection with PRP injection in the treatment for Plantar Fasciitis. Participants will be randomized in a 1:1 ratio, and assigned to steroid injection and PRP injection group through computer generated block randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (PRP) group (Experimental): The PRP will be prepared based on the Sengodan et al, 2020 study.
  Interventions: Drug: Platelet Rich Plasma (PRP) group
- Steroid group (Active Comparator): Steroid group will be treated with steroid injection. In this group, 2ml of Inj. Depo-Medrol 80 mg (Methylprednisolone) along with 1 ml lignocaine (0.25%) will be loaded in 5cc syringe and then the cocktail will be injected into medial calcaneal tuberosity at the most tender point using an aseptic technique as mentioned by Nishanth et.at,2018.
  After the procedure, participants will be advised not to involve in any kind of rigorous activity with the affected foot for at least two days and then gradually return to their regular activities. All patients will be counseled to follow up in the next visit at 3 months and 6 months. The end-line information will be again recorded at 3 months and 6 months.
  Interventions: Drug: Platelet Rich Plasma (PRP) group

INTERVENTIONS:
Drug: Platelet Rich Plasma (PRP) group — Platelet Rich Plasma (PRP) group will be intervened with PRP injection. The collection of 30 ml blood of patients into acid citrate dextrose tube under aseptic condition will be done and subjected for centrifugation at 2000 rpm (soft spin) through digital centrifuge machine speed control (REMI, R-8C PLUS). There will be three layers of blood, among them the supernatant layer and buff coat of plasma will be again subjected to centrifuge at 3000 rpm (hard spin). The upper two thirds of the tube containing platelet poor plasma will be discarded and finally, the lower one third concentrated platelet plasma superficial buffy coat will be injected into medial calcaneal tuberosity at the most tender point.
  Other Names: PRP intervention

SUMMARY:
Plantar fasciitis (PF) is the one of the most common orthopaedic problem resulting in heel pain. Previous evidence suggests that Platelet Rich Plasma (PRP) injection has better outcome in the long run as compared to the local steroid injection (SI). Although over the past many years, steroid injection was considered as the choice of treatment after the failure of conservative treatment methods, PRP therapy has shown promising results in the treatment of plantar fasciitis now-a-days. The aim of this study is to assess the effect of PRP injection compared with Steroid injection in the treatment of Plantar Fasciitis.

A hospital-based randomized clinical trial study will be carried out to compare the efficacy of the therapeutic effect between steroid injection and Platelet Rich Plasma injection in plantar fasciitis. A representative sample size of 78 patients aged 18 years to 60 years suffering from plantar fasciitis with failed conservative treatment will be intervened. The American Orthopedic Foot and Ankle Society (AOFAS) and the visual analog scale (VAS) scoring system will be recorded pre- and post-injection phases at 3 months and 6 months period. Statistical analyses will be performed using independent t-test and Mann Whitney U test to compare between the two means. The outcome of this study will help to guide the physicians to choose the better therapeutic approach among the patients suffering from plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis is a common and degenerative condition of plantar fascia resulting from excessive strain and micro-trauma on the planter surface of the foot. The prevalence of Plantar Fasciitis is estimated up to 7% in the general population and is common cause of plantar heel pain. The incidence of calcaneum spur with heel pain in the age group of 40 to 50 years is around 59% in the case of India. Plantar fasciitis is defined as localized inflammation and degeneration of the plantar aponeurosis, and it is the most common reason for presentation. Plantar Fasciitis is considered to be a self-limiting disease which resolves, in 80% to 90% of cases, within 10 months. This disease is very problematic for both doctors and patients. The majority of treatment options are non-surgical approaches due to the nature of the disease. The NSAIDS, shoe insert, stretching exercise or extracorporeal shockwave therapy are the common non-surgical therapy. Typically, these types of non-operative treatment are successful up to 90% of the patients with the condition and, in those patients who do not respond to non-operative treatment, injection therapies may be utilized.

The occurrence of plantar fasciitis is multifactorial. The risk factors may be extrinsic or intrinsic. Whatever may be the cause of plantar fasciitis, it is painful and affects the daily functioning of life. Orchard (2012) mentions the lifetime prevalence of plantar fasciitis as 10%, and it mostly affects the people aged 40 to 60 years, having no discrimination in gender. The prevalence of plantar fasciitis is estimated up to 7 % in general population. Goweda et al, 2015 found the prevalence of plantar fasciitis in Saudi Arabia as 57.8%. The number of cases of heel pain is increasing day by in Nepal. The prevalence of Plantar Fasciitis in Nepal could not be traced because of the lack of study in our population. However, different studies have been found in other perspectives. Different modalities of the treatment for PF are available. They are stretching exercise, soft heel pad shoe, ultrasound therapy, NSAIDs etc. If conservative treatment fails, the steroid injection is the preferred choice for the clinicians in practice, but this treatment has certain limitations as it can only reduce pain for a few months but not thereafter. Many studies suggest PRP treatment is more safe and beneficial than steroid injection in this manner. PRP therapy has been gaining popularity over the steroid therapy in the western world. But there are no studies done so far in the context of Nepal. Hence, this study will generate the empirical evidence to fill the knowledge gap for the treatment of PF.

ELIGIBILITY:
Inclusion Criteria:

* The patients having the pain over the plantar aspect of foot for more than 6 weeks with tenderness on palpation over the medial calcaneal tuberosity, failure of conservative treatment with physiotherapy, splints and NSAIDs.

Exclusion Criteria:

* Lumbar radiculopathy
* Existing trauma, previous surgery or any local pathology over the foot
* Patient on aspirin
* Bleeding disorders with low platelet counts
* Systemic disease like diabetes and rheumatoid arthritis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction | Six months
  Visual analog scale (VAS) will be used to measure the pain assessment at the three months and six months follow-up.
Functional mobility of the patients | Six months
  American Foot and Ankle Score (AFAS) ankle-Hindfoot scale will be used to measure the functional outcome of the patients at the three months and six months follow-up.

SECONDARY OUTCOMES:
Plantar fascia thickness | Six months
  Measure the changes of plantar fascia thickness in steroid injection and Platelet-Rich Plasma injection using ultrasonogram at six months

CONTACTS AND LOCATIONS:
Overall Officials: Rachit Sharma, MBBS, MS, Study Director — Nepal Orthopedic Hospital
Locations (1):
- Dev Ram Sunuwar, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lareau CR, Sawyer GA, Wang JH, DiGiovanni CW. Plantar and medial heel pain: diagnosis and management. J Am Acad Orthop Surg. 2014 Jun;22(6):372-80. doi: 10.5435/JAAOS-22-06-372. PMID 24860133
- [Result] Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. No abstract available. PMID 15152061
- [Result] League AC. Current concepts review: plantar fasciitis. Foot Ankle Int. 2008 Mar;29(3):358-66. doi: 10.3113/FAI.2008.0358. No abstract available. PMID 18348838
- [Result] Davis PF, Severud E, Baxter DE. Painful heel syndrome: results of nonoperative treatment. Foot Ankle Int. 1994 Oct;15(10):531-5. doi: 10.1177/107110079401501002. PMID 7834059
- [Result] Healey K, Chen K. Plantar fasciitis: current diagnostic modalities and treatments. Clin Podiatr Med Surg. 2010 Jul;27(3):369-80. doi: 10.1016/j.cpm.2010.03.002. Epub 2010 May 14. PMID 20691370
- [Result] Acevedo JI, Beskin JL. Complications of plantar fascia rupture associated with corticosteroid injection. Foot Ankle Int. 1998 Feb;19(2):91-7. doi: 10.1177/107110079801900207. PMID 9498581
- [Result] David JA, Sankarapandian V, Christopher PR, Chatterjee A, Macaden AS. Injected corticosteroids for treating plantar heel pain in adults. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009348. doi: 10.1002/14651858.CD009348.pub2. PMID 28602048
- [Result] Zhang JY, Fabricant PD, Ishmael CR, Wang JC, Petrigliano FA, Jones KJ. Utilization of Platelet-Rich Plasma for Musculoskeletal Injuries: An Analysis of Current Treatment Trends in the United States. Orthop J Sports Med. 2016 Dec 21;4(12):2325967116676241. doi: 10.1177/2325967116676241. eCollection 2016 Dec. PMID 28210648
- [Result] Baksh N, Hannon CP, Murawski CD, Smyth NA, Kennedy JG. Platelet-rich plasma in tendon models: a systematic review of basic science literature. Arthroscopy. 2013 Mar;29(3):596-607. doi: 10.1016/j.arthro.2012.10.025. Epub 2013 Jan 24. PMID 23352397
- [Result] Orchard J. Plantar fasciitis. BMJ. 2012 Oct 10;345:e6603. doi: 10.1136/bmj.e6603. No abstract available. PMID 23054045
- [Result] Say F, Gurler D, Inkaya E, Bulbul M. Comparison of platelet-rich plasma and steroid injection in the treatment of plantar fasciitis. Acta Orthop Traumatol Turc. 2014;48(6):667-72. doi: 10.3944/AOTT.2014.13.0142. PMID 25637732
- [Result] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Result] Jain K, Murphy PN, Clough TM. Platelet rich plasma versus corticosteroid injection for plantar fasciitis: A comparative study. Foot (Edinb). 2015 Dec;25(4):235-7. doi: 10.1016/j.foot.2015.08.006. Epub 2015 Aug 22. PMID 26362235
- [Derived] Sharma R, Chaudhary NK, Karki M, Sunuwar DR, Singh DR, Pradhan PMS, Gyawali P, Duwal Shrestha SK, Bhandari KK. Effect of platelet-rich plasma versus steroid injection in plantar fasciitis: a randomized clinical trial. BMC Musculoskelet Disord. 2023 Mar 7;24(1):172. doi: 10.1186/s12891-023-06277-1. PMID 36882804